CLINICAL TRIAL: NCT01094730
Title: A Multi-site Dispensing Evaluation Comparing a New Galyfilcon A Prototype Lens With a Marketed Galyfilcon A Contact Lens
Brief Title: Pilot Evaluation of a New Galyfilcon A Contact Lens Compared to a Marketed Galyfilcon A Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-1636AY
Record Dates: First submitted 2010-03-24; First posted 2010-03-29 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- galyfilcon A prototype/marketed galyfilcon A (Other): The galyfilcon A prototype lens worn daily for 12-16 days during the first period then the marketed galyfilcon A lens worn daily for 12-16 days during the second period.
  Interventions: Device: galyfilcon A prototype lens; Device: marketed galyfilcon A lens
- marketed galyfilcon A/galyfilcon A prototype (Other): The marketed galyfilcon A lens worn daily for 12-16 days during the first period then the galyfilcon A prototype lens worn daily for 12-16 days during the second period; during each period.
  Interventions: Device: galyfilcon A prototype lens; Device: marketed galyfilcon A lens

INTERVENTIONS:
Device: galyfilcon A prototype lens — Experimental silicone hydrogel contact lens
Device: marketed galyfilcon A lens — Marketed silicone hydrogel contact lens.
  Other Names: ACUVUE(R) ADVANCE(TM)

SUMMARY:
The purpose of this study is to compare lens surface characteristics and comfort between an experimental contact lens and a marketed contact lens.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 18 years of age and no more than 39 years of age.
* The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of daily wear (DW) for a minimum of 1 month prior to the study) and willing to wear the study lenses on a daily wear basis (defined as a minimum of 6 hours of wear per day at least five days of the week) for the duration of the study.
* The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and - 9.00D.
* Any cylinder power must be ≤ -0.75D.
* The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
* The subject must read and sign the Statement of Informed Consent.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

* Ocular or systemic allergies or disease which might interfere with contact lens wear.
* Systemic disease or use of medication which might interfere with contact lens wear.
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
* Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Pregnancy or lactation.
* Diabetes.
* Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
* Habitual contact lens type is toric, multifocal, or is worn as extended wear.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-04-01 (Actual); Study Completion 2010-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Cupertino, California
  - Huntington Beach, California
  - Los Angeles, California
  - Pismo Beach, California
  - Jacksonville, Florida
  - Orlando, Florida
  - East Lansing, Michigan
  - Columbus, Ohio
  - Amarillo, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were five subjects enrolled who were not randomized to a study arm due to exclusion criteria dropping the study enrollment from 185 to 180.
Groups:
- Galyfilcon A Prototype/Marketed Galyfilcon A: The galyfilcon A prototype lens worn daily for 12-16 days during the first period then marketed galyfilcon A lens worn daily for 12-16 days during the second period.
- Marketed Galyfilcon A/Galyfilcon A Prototype: The marketed galyfilcon A lens worn daily for 12-16 days during the first period then the galyfilcon A prototype lens worn daily for 12-16 days during the second period.
Period: Period 1 (14 Days)
Arm/Group | Galyfilcon A Prototype/Marketed Galyfilcon A | Marketed Galyfilcon A/Galyfilcon A Prototype
Started | 92 | 88
Completed | 90 | 86
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — No time for the follow-up visit | 1 | 0
Not completed — Unsatisfactory visual response | 1 | 0
Period: Period 2 (14 Days)
Arm/Group | Galyfilcon A Prototype/Marketed Galyfilcon A | Marketed Galyfilcon A/Galyfilcon A Prototype
Started | 90 | 86
Completed | 87 | 84
Not Completed | 3 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — No time for the follow-up visit | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Unsatisfactory lens fitting | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline summary was conducted on all enrolled subjects who have the demographic data. Two enrolled subjects were excluded from the Baseline summary for age and gender categories due to missing demographic data, reducing the count from 185 to 183; one subject was ineligible and the other one withdrew their consent.
Groups:
- All Subjects: All enrolled subjects who have the demographic data and worn at least one study lens.
Arm/Group | All Subjects
Number analyzed (Participants) | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (5.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 55
Region of Enrollment [Number; unit: participants]
  United States | 183

OUTCOME MEASURES:

1. Primary Outcome: Lens Front Surface Deposits at Day 7
Description: Deposits on the front surface of each lens were examined by the investigator after 7 days of lens wear, and graded on a 5-point scale; 0 = no deposit, 1 = 1%-5% deposits, 2 = 6%-15% deposits, 3 = 16%-25% deposits, and 4 = 25% or more deposits. The grades were categorized into binary variable: grade 0 or 1 Vs. grade 2 or higher.
Time Frame: Evaluated at Day 7
Population: Analysis was conducted on subjects who successfully completed the study.
Measure: Mean (Standard Deviation); unit: dichotomized grading scale
Units Other Than Participants: eyes
Arm/Group | Galyfilcon A Prototype Lens | Marketed Galyfilcon A Lens
Number analyzed (Participants) | 171 | 169
Number analyzed (eyes) | 341 | 338
dichotomized grading scale | 1.53 (0.769) | 1.53 (0.715)

2. Secondary Outcome: Subject Reported Overall Lens Comfort at Day 7
Description: The overall lens comfort was assessed at Day 7 using the Contact Lens User Experience (CLUE) questionnaire. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging)in a contact lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable /positive response. 97% of the scores fall within 0 and 120 (mean +/-3*SD).
Time Frame: Evaluated at Day 7
Population: Analysis was conducted on subjects who successfully completed the study.
Measure: Mean (Standard Error); unit: CLUE points
Groups:
- Galyfilcon A Prototype Lens: Experimental silicon hydrogel contact lens.
- Marketed Galyfilcon A Lens: Marketed silicon hydrogel contact lens.
Arm/Group | Galyfilcon A Prototype Lens | Marketed Galyfilcon A Lens
Number analyzed (Participants) | 170 | 170
CLUE points | 60.7787 (2.3993) | 59.3206 (2.3850)

3. Primary Outcome: Lens Front Surface Deposits at Day 14
Description: Deposits on the front surface of each lens were examined by the investigator after 14 days of lens wear, and graded on a 5-point scale; 0 = 0% deposits, 1 = 1%-5% deposits, 2 = 6%-15% deposits, 3=16%-25% deposits, and 4= 25% or more deposits. The grades were categorized into binary variable: grade 0 or 1 vs. grade 2 or higher.
Time Frame: Evaluated at Day 14
Population: Analysis was conducted on subjects who successfully completed the study.
Measure: Mean (Standard Deviation); unit: dichtomized grading scale
Units Other Than Participants: Contact Lenses
Arm/Group | Galyfilcon A Prototype Lens | Marketed Galyfilcon A Lens
Number analyzed (Participants) | 169 | 170
Number analyzed (Contact Lenses) | 338 | 340
dichtomized grading scale | 1.61 (0.681) | 1.67 (0.759)

4. Secondary Outcome: Subject Reported Overall Lens Comfort at Day 14
Description: The overall lens comfort was assessed at Day 14 using the CLUE questionnaire. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging)in a contact lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable /positive response. 97% of the scores fall within 0 and 120 (mean +/-3*SD).
Time Frame: Evaluated at Day 14
Population: Analysis was conducted on subjects who successfully completed the study.
Measure: Mean (Standard Error); unit: CLUE points
Arm/Group | Galyfilcon A Prototype Lens | Marketed Galyfilcon A Lens
Number analyzed (Participants) | 169 | 169
CLUE points | 57.3230 (2.4790) | 55.4675 (2.4694)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded when the subjects were exposed to the Investigational lenses.
Groups:
- All Subjects: All subjects were to wear both lenses during the course of the study.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/181
Other Adverse Events (participants affected / at risk) | 0/181

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires the agreement and written authorization of the Sponsor.